CLINICAL TRIAL: NCT00728013
Title: China Intensive Lipid Lowering With Statins in Acute Coronary Syndrome
Acronym: CHILLAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Yong Huo, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006BAI01A02-12
Record Dates: First submitted 2008-07-29; First posted 2008-08-05 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; intensive lipid-lowering; statins
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): intensive statin group
  Interventions: Drug: Atorvastatin
- B (Experimental): moderate statin group
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Eligible patients are randomly assigned (1:1 ratio) by center to intensive statin therapy (atorvastatin, 20 or 40 mg/d, or equivalent dose of other statins)
  Arms: A
Drug: Atorvastatin — Eligible patients are randomly assigned (1:1 ratio) by center to moderate therapy (atorvastatin, 10 mg/d, or equivalent dose of other statins).
  Arms: B

SUMMARY:
In summary, the CHILLAS study will be the first multicenter study performed in a Chinese population using a patient-level analysis to compare the effects and safety of intensive statin therapy with that of moderate statin therapy. Therefore, it will determine whether "lower is better", that is, whether LDL cholesterol lowering to a level of approximately 100mg/dl provides a benefit inferior to that of LDL cholesterol lowering to a much lower level; examine the role of inflammatory markers in predicting cardiac events and response to statin therapy; and evaluate the effects of statin therapy on regression of coronary atherosclerosis using IVUS.

DETAILED DESCRIPTION:
The CHILLAS study is planned to evaluate whether intensive treatment with statins for 2 years results in a reduction of cardiovascular events in patients with ACS. A total of 1,600 patients will be randomly assigned to receive intensive statin therapy (atorvastatin, 20 or 40 mg/d, or equivalent dose of other statins) or moderate therapy (atorvastatin, 10 mg/d, or equivalent dose of other statins). Both groups receive dietary counseling. Over a 2-year follow-up period, the primary outcome measure is the time to occurrence of cardiac death, nonfatal acute myocardial infarction, revascularization with either percutaneous coronary intervention or coronary-artery bypass grafting, documented unstable angina or severe heart failure requiring emergency hospitalization, and stroke. The planned duration is between December 2006 and December 2009.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute coronary syndrome
* Clinically stable for 24 hours

Exclusion Criteria:

* Hypersensitive to statins
* Receiving therapy with atorvastatin at a dose greater than 20 mg per day before enrollment or lipid-lowering therapy with fibric acid derivatives or niacin that can not be discontinued
* Having a coexisting condition that shortened expected survival to less than two years
* Having obstructive hepatobiliary disease or other serious hepatic or kidney disease
* Having an unexplained elevation in the creatine kinase level that was more than three times the upper limit of normal and that was not related to myocardial infarction
* Having undergone surgery or serious trauma within the preceding two months
* Having been in the final stage of chronic congestive heart failure
* Having a baseline level of LDL cholesterol less than 50mg/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac death, nonfatal AMI, revascularization with either percutaneous coronary intervention or coronary-artery bypass grafting, documented unstable angina or severe heart failure requiring emergency rehospitalization, and stroke | 2 years

SECONDARY OUTCOMES:
The secondary endpoints include total mortality | 2 years
LDL cholesterol success rate | 2 years
Percentage rate of plaque regression | 2 years
In addition, changes in CRP from baseline to specified measurement time points will be calculated | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shuiping Zhao, MD, Study Director — Ministry of Education of the People's Republic of China
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China